CLINICAL TRIAL: NCT04617327
Title: Short Course Pre-operative RadiothErapy for Soft Tissue SarcOmas - a Phase I/II Trial (PRESTO)
Brief Title: Pre-operative RadiothErapy for Soft Tissue SarcOmas
Acronym: PRESTO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Fabio Cury, Principal Investigator/Radiation Oncologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MUHC-RIMUHC
Record Dates: First submitted 2020-06-25; First posted 2020-11-05 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Soft Tissue Sarcoma Adult
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental : Short Course Pre-operative RadiothErapy (Experimental): As part of the planning process, you need to undergo a CT Simulation.It is special type of CT scan used to measure and design the radiation fields to precisely target the tumor.It is done at the Radiation Oncology Department at the MUHC. Some patients may be asked to also undergo an MRI Simulation, and the CT simulation. You may asked to provide a blood sample to ensure good kidney function prior to the CT and MRI scans. Both CT and MRI simulations are considered standard of care.
  Once the simulation studies are done, there is about a 2 week waiting period for radiation planning prior to starting the radiation treatments.
  The hypofractionation technique will be delivering five fractions (one fraction delivered every 2nd day) of 7 Gy daily of external beam radiotherapy (EBRT) over a period of one and half weeks for a total of 35 Gy. The treatment should last approximately 30 minutes. Once treatments are done, there is a 4 to 6 week wait for surgery.
  Interventions: Radiation: Hypofractionation

INTERVENTIONS:
Radiation: Hypofractionation — Shorter radiation therapy means that a higher dose will be given on a daily basis. The goal is to target microscopic disease and decrease the chances of local recurrence.
  Organs at risk (OAR) will receive doses following the constraints from the Timmerman tables used for reference when using 5 or more fractions of EBRT.
  Treatment will be delivered every 2nd day, for a maximum of 3 fractions per week. Daily pretreatment Image Guided Radiotherapy Images (IGRT) (Cone-Beam CT - CBCT) will be co-registered with the CT simulation dataset to adjust patient position before each treatment by matching the bone adjacent to the planned tumour volume (PTV). Treatment will be administered if there is <3 mm in any dimension, or rotation is <3 degrees. If the isocentre set-up exceeds 3 mm at any given treatment session, the treatment couch will be translated to restore its planned position.
  Other Names: Hypofractionated Radiation Therapy

SUMMARY:
Soft tissue sarcomas (STSs) are malignant tumours that arise in any of the mesodermal tissues in the body including muscles, fibrous tissues, bone and cartilage, adipose tissue, and blood vessels, most frequently in the extremities (40%), trunk and retroperitoneum (40%).

Traditionally, the prescription schedule for conventional preoperative RT is a regimen of 50 Gy in fractions of 1.8-2 Gy per day. Concerns regarding this regimen include the delay to definitive surgery and the higher rate of wound complications compared to post-operative radiotherapy. Hypofractionated RT is a prescription schedule in which the total dose of radiation is delivered in larger doses per fraction in fewer fractions allowing the delivery of a higher biologically effective dose (BED) to the tumour than with conventional RT [7] during a shorter period of time.

DETAILED DESCRIPTION:
This will be a phase I/II study of hypofractionation delivering five fractions (one fraction delivered every 2nd day) of 7 Gy of external beam radiotherapy over 5 fractions (one and half week period) in patients with localized STSs who are planned to receive pre-operative radiotherapy. Patients will undergo surgery 4-6 weeks after completion of RT.

Pre-treatment evaluation will be according to standard practice:

History and Physical Exam

* height,
* weight
* history (diabetes, vascular disease)

Radiology

* MRI of primary site or
* CT if MRI not tolerated
* CT chest

Quality of Life

* Musculoskeletal Tumour Society Rating Scale
* Toronto Extremity Salvage Score (TESS)

Follow-up assessment will be done as follows:

History and Physical Exam

* Acute radiation toxicity
* During RT and 2 weeks after end of RT

Acute surgical toxicity - wound assessment

* At hospital discharge,
* 2 weeks post-surgery
* 1 month post-surgery
* 3 months post-surgery
* 6 months post-surgery

Late toxicity (skin, subcutaneous, bone, joint) & peripheral limb edema

- Every 6 months thereafter

Radiology

* Chest CT-scan
* Within 1 month pre-surgery
* Standard thereafter

MRI or CT scan of primary site

* Prior to surgery, as standard
* Every 3-6 months or as needed after surgery

Quality of life Questionnaires

* Toronto Extremity Salvage Score (TESS
* Musclo Tumor Rating Scale (MSTS)
* At months 1,3,6, 12, 18 and 24 after surgery.
* Yearly thereafter up to 5 years

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven STS of the extremities, above the knee, or trunk following review by our pathologist

  * Lesions smaller than 15cm in largest dimension
  * Deemed appropriate for preoperative radiotherapy and conservative surgery following patient assessment by a radiation oncologist and surgical oncologist
  * Lesion is primary or locally recurrent. Patients who underwent unplanned non-oncological excision ("whoops" procedure) at a referring hospital are NOT eligible
  * No previous radiation therapy
  * ECOG 0-2 (or Karnofsky Performance Status ≥ 70) within 60 days prior to registration
  * Resectable primary lesion with or without distant metastasis
  * Age ≥ 18
  * Patient must be able to provide study-specific informed consent prior to study entry
  * Patient is available for treatment and follow-up

Exclusion Criteria:

* Patients who underwent unplanned non-oncological excision ("whoops" procedure) at a referring hospital

  * Lesions below the knee
  * Prior or concurrent invasive malignancy (except non-melanomatous skin cancer) or lymphomatous/hematogenous malignancy, unless continually disease free for a minimum of 5 years
  * Regional lymph node involvement
  * Previous irradiation to the area to be treated
  * Other major medical illness deemed to preclude safe administration of protocol treatment or required follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute RadiationToxicity using Common Terminology Criteria for Adverse Events (CTCAE) V.5 | 1 month
  To assess, skin reactions and wound healing

SECONDARY OUTCOMES:
Physicians Muscle Tumor Rating Scale | 1 year
  To assess the amount of difficulty performing activities, including motion, strength and stability

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Cury, MD, Principal Investigator — Research Institute of McGill University Health Centre
Locations (1):
- McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec, Canada